CLINICAL TRIAL: NCT00201526
Title: Bipolar Research And Innovation Network - BRAIN
Status: Recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Other Study IDs: 10671
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: RCT
- Control group: RCT

SUMMARY:
To describe the broad spectrum of Bipolar Disorder patients admitted to out-patient and in-patient psychiatric departments in Norway. Include all admitted Bipolar patients both with and without co-morbid disorders.

DETAILED DESCRIPTION:
Norway is both social, genetically and culturally a homogeneous society. The health service is public and has a nearly total responsibility for psychiatric care in given catchment areas. This provides excellent opportunities to describe the frequencies and patterns of the broad spectrum of bipolar illness, including co-morbid substance use disorders, to follow the patients for several years and to do molecular genetic mapping.

Methods: Participating centers consist of outpatient clinics and hospital departments from different parts of Norway and one third-line clinic with referrals from all over Norway. Specifically trained clinicians in each center include bipolar patients systematically and perform the patient evaluation as part of their clinical duties. In addition, CT or MRI scans and EEG are performed and blood samples are collected for clinical chemistry screening and for DNA sampling.

ELIGIBILITY:
Inclusion Criteria:

* All admitted patients giving written consent to participate in the study

Exclusion Criteria:

* Patients without competence for consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Secondary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2003-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Difference in remission | 15 years
  Clinical Interview. Difference (MADRES) in remission between the study and control group.
Difference in response | 15 years
  Clinical Interview. Difference (MADRS) in response between the study and control group.

SECONDARY OUTCOMES:
GAF | 15 years
  Clinical Interview. Global Assessment of Function
Current and concomitant medication | 1 year
  Clinical Interview.
SF36 | 1 year
  Clinical Interview.
MADRS | 1 year
  Clinical Interview.
IDS Inventory of depressive sympthoms | 1 year
  Clinical Interview.
CGI-BP Clinical Global Index - Bipolar | 1 year
  Clinical Interview.
PGI-1 (Patient global index) | 1 year
  Clinical Interview.
YMRS (Young mania rating scale) | 1 year
  Clinical Interview.
MSIF (Quality of life scale) | 1 year
  Clinical Interview.
MMS (Minimal mental scale) | 1 year
  Clinical Interview.
EMQ (Neuropsychology) | 1 year
  Clinical Interview.
UKU (Medication side effects) | 1 year
  Clinical Interview.
SAE-form (Serious adverse events) | 1 year
  Clinical Interview.
Cytokines | 1 year
  Laboratory
Cortisol | 1 year
  Laboratory
Substance used | 1 st week
  Laboratory, Urine
Compliance (medication) | 1 st year
  Clinical interview
TEMPS-A (Temperament) | Week 26
  Clinical interview
Migraine (Clinical interview) | Week 1 and week 26
  Clinical interview

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Morken, PhD MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Medical Faculty, Norwegian University of Science And Technology, Trondheim, Norway

REFERENCES:
- [Background] Kessler U, Vaaler AE, Schoyen H, Oedegaard KJ, Bergsholm P, Andreassen OA, Malt UF, Morken G. The study protocol of the Norwegian randomized controlled trial of electroconvulsive therapy in treatment resistant depression in bipolar disorder. BMC Psychiatry. 2010 Feb 23;10:16. doi: 10.1186/1471-244X-10-16. PMID 20178636
- [Background] Kessler U, Schoeyen HK, Andreassen OA, Eide GE, Hammar A, Malt UF, Oedegaard KJ, Morken G, Sundet K, Vaaler AE. Neurocognitive profiles in treatment-resistant bipolar I and bipolar II disorder depression. BMC Psychiatry. 2013 Apr 4;13:105. doi: 10.1186/1471-244X-13-105. PMID 23557429
- [Background] Kessler U, Schoeyen HK, Andreassen OA, Eide GE, Malt UF, Oedegaard KJ, Morken G, Sundet K, Vaaler AE. The effect of electroconvulsive therapy on neurocognitive function in treatment-resistant bipolar disorder depression. J Clin Psychiatry. 2014 Nov;75(11):e1306-13. doi: 10.4088/JCP.13m08960. PMID 25470096
- [Background] Schoeyen HK, Kessler U, Andreassen OA, Auestad BH, Bergsholm P, Malt UF, Morken G, Oedegaard KJ, Vaaler A. Treatment-resistant bipolar depression: a randomized controlled trial of electroconvulsive therapy versus algorithm-based pharmacological treatment. Am J Psychiatry. 2015 Jan;172(1):41-51. doi: 10.1176/appi.ajp.2014.13111517. Epub 2014 Oct 31. PMID 25219389
- [Background] Bjoerke-Bertheussen J, Schoeyen H, Andreassen OA, Malt UF, Oedegaard KJ, Morken G, Sundet K, Vaaler AE, Auestad B, Kessler U. Right unilateral electroconvulsive therapy does not cause more cognitive impairment than pharmacologic treatment in treatment-resistant bipolar depression: A 6-month randomized controlled trial follow-up study. Bipolar Disord. 2018 Sep;20(6):531-538. doi: 10.1111/bdi.12594. Epub 2017 Dec 21. PMID 29267990
- [Derived] Drange OK, Saether SG, Finseth PI, Morken G, Vaaler AE, Arntsen V, Henning O, Andreassen OA, Elvsashagen T, Malt UF, Boen E. Differences in course of illness between patients with bipolar II disorder with and without epileptiform discharges or other sharp activity on electroencephalograms: a cross-sectional study. BMC Psychiatry. 2020 Dec 7;20(1):582. doi: 10.1186/s12888-020-02968-4. PMID 33287748
- [Derived] Drange OK, Vaaler AE, Morken G, Andreassen OA, Malt UF, Finseth PI. Clinical characteristics of patients with bipolar disorder and premorbid traumatic brain injury: a cross-sectional study. Int J Bipolar Disord. 2018 Sep 10;6(1):19. doi: 10.1186/s40345-018-0128-6. PMID 30198055